CLINICAL TRIAL: NCT05502120
Title: A Comparison of Visualization of the Larynx With the Vie Scope Versus Standard Macintosh Laryngoscope in Morbidly Obese Patients.
Brief Title: A Comparison of Vie-Scope and Macintosh Blade Laryngoscopes in Morbidly Obese.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RNN/49/21/KB
Record Dates: First submitted 2022-06-22; First posted 2022-08-16 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-06

CONDITIONS: Obesity, Morbid; Intubation Complication
Keywords: morbid obesity; endotracheal intubation
MeSH Terms: conditions — Obesity, Morbid | interventions — Laryngoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macintosh blade (Active Comparator): Visualisation of entrance to larynx using Standard Macintosh blade laryngoscope followed by Visualisation of entrance to larynx using Vie-Scope laryngoscope
  Interventions: Device: Laryngoscopy with Macintosh blade laryngoscope
- Vie-Scope (Experimental): Visualisation of entrance to larynx using Vie-Scope laryngoscope after visualisation using Macintosh blade laryngoscope
  Interventions: Device: Laryngoscopy with Vie-Scope laryngoscope

INTERVENTIONS:
Device: Laryngoscopy with Vie-Scope laryngoscope — Evaluation of laryngeal view using Vie-Scope laryngoscope, intubation efficacy, complications
  Arms: Vie-Scope
Device: Laryngoscopy with Macintosh blade laryngoscope — Evaluation of laryngeal view using stnadard Macintosh blade laryngoscope
  Arms: Macintosh blade

SUMMARY:
Macintosh laryngoscope is still considered a standard for tracheal intubation, however, visualization of the glottis may be inadequate mainly in morbidly obese patients. The Vie Scope is a novel type of laryngoscope consisting of a straight, shielded, illuminated tube that offers intubation via a bougie using the paraglossal technique. In this prospective, non-randomized study, we tested the research hypothesis that the use of Vie Scope may improve visualization of the larynx in comparison with the Macintosh blade.

DETAILED DESCRIPTION:
Prior to tracheal intubation, all patients were placed in the head-elevated laryngoscopy position (HELP). All study subjects were anesthetized with the concordance to European Society for Peri-Operative Care of Obese Patient (www.espcop.eu) protocols: proper positioning, pre-oxygenation with CPAP, induction of anesthesia with propofol 2.0 mg kg-1 of corrected body weight; for muscle relaxation rocuronium 0.6 mg kg-1 of ideal body weight (IBW); ketamine 50 mg ; lidocaine 100 mg, and fentanyl 0.1 mg. After achieving 100% neuromuscular block confirmed by TOF-Watch monitoring, laryngoscopy was performed by the anesthesiologist familiar with the use of both Vie Scope and Macintosh blade laryngoscope, and also experienced in bariatric anesthesia. All anesthesiologists participating in the study underwent training with Vie Scope on the manikin model.

The evaluation of glottis visualization in direct laryngoscopy using Cormack-Lehane scale (CL) in all patients was performed in sequence using two laryngoscopes: first Macintosh blade laryngoscope (MCL) and then Vie Scope laryngoscope (VS). Tracheal intubation was performed with the VS. The study subjects all received oxygen using nasal CPAP in order to maintain sufficient oxygenation

ELIGIBILITY:
Inclusion Criteria:

* morbid obesity BMI>40 kg/m2
* scheduled for elective bariatric procedure
* no anatomy abnormalities of upper airway

Exclusion Criteria:

* lack of conscent
* predicted difficult intubation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Improvement in laryngeal view | through study completion, an average of 1 year
  Expected improvement in laryngeal view obtained with the use of Vie-Scope laryngoscope

SECONDARY OUTCOMES:
intubation efficiency | through study completion, an average of 1 year
  Success of intubation using Vie-Scope laryngoscope

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No